CLINICAL TRIAL: NCT05817461
Title: An Open-Label, Two-Part Sequential Study Designed to Assess the Mass Balance Recovery, Absorption, Metabolism, Excretion of [14C]AZD0780 and the Absolute Bioavailability of AZD0780 in Healthy Male Subjects
Brief Title: An ADME Study of [14C]AZD0780 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7960C00004
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Dyslipidaemia
MeSH Terms: conditions — Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD0780 (Experimental): In Part 1, one oral dose of AZD0780 and one intravenous dose of [14C]AZD0780. In Part 2, one oral dose of [14C]AZD0780
  Interventions: Drug: AZD0780 tablet; Drug: [14C]AZD0780 Solution for Infusion; Drug: [14C]AZD0780 Oral Solution

INTERVENTIONS:
Drug: AZD0780 tablet — oral, fasted
  Other Names: AZD0780
Drug: [14C]AZD0780 Solution for Infusion — intravenous
  Other Names: [14C]AZD0780
Drug: [14C]AZD0780 Oral Solution — oral, fasted
  Other Names: [14C]AZD0780

SUMMARY:
The Sponsor is developing a new test medicine, AZD0780, with the aim to lower low-density lipoprotein cholesterol (LDL-C, fatty deposits) levels and cardiovascular (heart disease) risk, when given on top of standard care.

This two-part healthy volunteer study will try to identify how the test medicine is taken up, broken down and removed from the body. To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14; also referred as 14C) which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

This study will take place at one non-NHS site, enrolling up to 8 male volunteers aged between 30 and 55 years.

DETAILED DESCRIPTION:
The Sponsor is developing a new test medicine, AZD0780, with the aim to lower low-density lipoprotein cholesterol (LDL-C, fatty deposits) levels and cardiovascular (heart disease) risk, when given on top of standard care. High levels of LDL-C can build up on the walls of blood vessels, forming plaques which can increase the risk of heart disease and stroke.

This two-part healthy volunteer study will try to identify how the test medicine is taken up, broken down and removed from the body.

To help investigate this, the test medicine is radiolabelled, which means that the test medicine has a radioactive component (carbon-14; also referred as 14C) which helps us to track where the test medicine is in the body. The safety and tolerability of the test medicine will also be studied.

This study will take place at one non-NHS site, enrolling up to 8 male volunteers aged between 30 and 55 years.

In Part 1, volunteers will receive a single oral dose of AZD0780 on Day 1. The volunteers will then receive a single intravenous dose of [14C]AZD0780, 2.25 hours after the oral dose. Volunteers will be discharged on Day 8. Following a minimum 14 day washout period, all volunteers who participated in Part 1 of the study will be admitted to the clinical unit for Part 2. In Part 2, the volunteers will receive a single oral dose of [14C]AZD0780 on Day 1. Volunteers will be discharged on Day 11, however, if relevant radioactivity criteria have not been met, volunteers may need to remain at the clinical unit until Day 13. If relevant criteria have not been met at this point, home collections of urine and/or faeces may be required.

Volunteers will receive a follow up phone call between Day 18 and 21.

Volunteer's blood and urine and faeces will be taken throughout the study for analysis of the test medicine and for their safety.

Volunteers are expected to be involved in this study for 10 weeks from screening to the follow up call.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Must be willing and able to communicate and participate in the whole study.
* Healthy male subjects aged 30 to 55 years inclusive at the time of signing informed consent.
* Must agree to adhere to the contraception requirements defined in the Clinical Protocol
* Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day).

Exclusion Criteria:

* History of any clinically significant disease or disorder (e.g. cardiovascular, pulmonary, GI, liver, renal, neurological, musculoskeletal ,endocrine, metabolic, malignant, psychiatric, major physical impairment, skin abnormalities and glucose metabolism abnormalities) which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of clinically significant GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0780. Hay fever is allowed unless it is active.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
* Evidence of current SARS-CoV-2 infection
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed.
* Clinically significant abnormal findings in vital signs, at screening or admission, as judged by the investigator.
* Clinically significant abnormalities on 12-lead ECG, at screening or admission, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), and human immunodeficiency virus (HIV) 1 and 2 antibody
* Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min using the Cockcroft-Gault equation
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer. Note: subjects consented and screened, but not randomised in this study or a previous Phase I study, are not excluded.
* Subjects who report to have previously received AZD0780.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
* Subjects who have been administered IMP in an ADME study in the last 12 months.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than 4 g of paracetamol/acetaminophen per day), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life. COVID-19 vaccines are accepted concomitant medications. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no PD activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardise the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks or 5 half-lives, whichever is longer, prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse in the past 2 years or excessive intake of alcohol (>21 units per week [1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type]) or as judged by the investigator.
* A confirmed positive alcohol breath test at screening or admission.
* Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.
* A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
* Confirmed positive drugs of abuse test result at screening or admission.
* Excessive intake of caffeine-containing drinks or food (e.g. coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g. >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Subjects with pregnant or lactating partners
* Planned in-patient surgery, dental procedure or hospitalisation during the study.
* Involvement of any Astra Zeneca, Quotient or study site employee or their close relatives.
* Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e. during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the investigator.
* Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) - Part 1 | Plasma sample collection from pre-dose to 168 hours post-dose
  Absolute bioavailability based on AUC0-inf of oral formulation compared to IV adjusted for dose
Area under the curve from time 0 extrapolated to infinity for AZD0780 and total radioactivity (AUC0-inf) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Time to maximum concentration (tmax) for AZD0780 and total radioactivity - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Maximum observed concentration (Cmax) for AZD0780 and total radioactivity - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Area under the curve from time 0 to the time of last measurable concentration for AZD0780 and total radioactivity (AUC0-t) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUCextrap) and total radioactivity - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Terminal elimination half-life for AZD0780 (t1/2) and total radioactivity - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD0780 (λz) and total radioactivity - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Total body clearance calculated after a single IV administration (CL) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single IV administration (Vz) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Volume of distribution at steady state after a single IV administration (Vss) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) - Part 1 | Plasma sample collection from pre-dose until 168 hours post-dose
  PK of AZD0780 and [14C]AZD0780 in plasma
Amount of AZD0780 excreted (Ae) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD0780 in urine and faecal samples
Amount of AZD0780 excreted expressed as a fraction of dose excreted (%Ae) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD0780 in urine and faecal samples
The cumulative amount of AZD0780 exreted (CumAe) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD0780 in urine and faecal samples
Cumulative amount of AZD0780 excreted expressed as a fraction of dose excreted (Cum%Ae) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  Mass balance of total radioactivity (TR) of [14C]AZD0780 in urine and faecal samples
Time to maximum concentration (tmax) for AZD0780 and total radioactivity - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Maximum observed concentration (Cmax) for AZD0780 and total radioactivity - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Area under the curve from time 0 to the time of last measurable concentration for AZD0780 and total radioactivity (AUC0-t) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Area under the curve from time 0 extrapolated to infinity for AZD0780 and total radioactivity (AUC0-inf) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUCextrap) and total radioactivity - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Terminal elimination half-life for AZD0780 (t1/2) and total radioactivity - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD0780 (λz) and total radioactivity - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Total body clearance calculated after a single extravascular administration where F (fraction of dose bioavailable) is unknown (CL/F) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Apparent volume of distribution based on the terminal phase calculated using AUC(0-inf) after a single extravascular administration where F (fraction of dose bioavailable) is unknown (Vz/F) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces
Renal clearance calculated using plasma AUC (CLR) - Part 2 | Urine and faecal samples collected from pre-dose until 240 hours post-dose
  PK of AZD0780 in urine and faeces

SECONDARY OUTCOMES:
Number of subjects with treatment-related adverse events - Part 1 and Part 2 | Through study duration, an average of 10 weeks
  To provide additional safety and tolerability information for AZD0780 by assessing the incidence of AEs
Blood:plasma concentration ratios - Part 2 | Whole blood samples and plasma samples collected from pre-dose until 240 hours post-dose
  Blood:plasma concentration ratios of total radioactivity
Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating TR (plasma) or accounting for 10% or more of the dose in urine and faeces - Part 2 | Plasma, urine and faecal samples collected from pre-dose until 240 hours post-dose
  Metabolite profiling and structural identification from plasma, urine and faecal samples.
  Metabolites are to be reported in a separate report after the Clinical Study Report is final.

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-DT.pharmacm.com/DT/Home

REFERENCES:
- See also: D7960C00004 CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7960C00004&attachmentIdentifier=290c0787-aa9e-4b1a-93ee-2809b2a3bcb0&fileName=d7960c00004-study-synopsis_Final_Redacted_18Apr2024.pdf&versionIdentifier=
- See also: Results posted on AZCT.com — https://www.astrazenecaclinicaltrials.com/study/D7960C00004/